CLINICAL TRIAL: NCT05475119
Title: Effect of High Flow Nasal Cannula (HFNC) Versus Continues Positive Airway Pressure (CPAP) in Adults With Obstructive Sleep Apnea
Brief Title: Effect of High Flow Nasal Cannula Versus Continues Positive Airway Pressure in Adults With Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Siraj Omar Wali, Director of Sleep Medicine and Research Center, Professor of Medicine, King Abdulaziz University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 724-19
Record Dates: First submitted 2022-06-22; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants diagnosed with Obstructive Sleep Apnea (Experimental): The participants will sleep three nights at the sleep lab and undergo in their first night, Polysomnography (PSG). Then at random, some of them will do CPAP titration in the second night followed by HFNC titration in the third night. While others will do HFNC titration in the second night followed by CPAP titration in the third night
  Interventions: Device: Continuous Positive Airway Pressure (CPAP); Device: High Flow Nasal Cannula (HFNC)

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) — Continuous Positive Airway Pressure (CPAP) is a form of positive airway pressure ventilation in which a constant level of pressure greater than atmospheric pressure is continuously applied to the upper respiratory tract of an individual.
Device: High Flow Nasal Cannula (HFNC) — High Flow Nasal Cannula (HFNC) is an oxygen supply system capable of delivering up to 100% humidified and heated oxygen at a flow rate of up to 60 liters per minute

SUMMARY:
The participants whom undergo Polysomnography study (Sleep study) and are found to have mild, moderate or severe Obstructive Sleep Apnea (OSA) will have two consecutive titration nights. Randomly, they'll do (CPAP) titration followed by (HFNC) titration or vice versa. To explore the possibility of the CPAP not being superior to HFNC in reduction of sleep apnea events.

DETAILED DESCRIPTION:
The participants undergo three nights in the Sleep Lab. In their first night they perpetrate Polysomnography study (Sleep study) and then classifies to have mild, moderate or severe Obstructive Sleep Apnea (OSA) or not. Those who are diagnosed with OSA, will undergo two consecutive titration nights. Randomly, they'll do (CPAP) titration followed by (HFNC) titration or vice versa. To explore the possibility of the CPAP not being superior to HFNC in reduction of sleep apnea events.

ELIGIBILITY:
Inclusion Criteria:

* Adults patient aging above 18 years
* Diagnosed with Obstructive Sleep Apnea (OSA) based on Polysomnography (PSG) ranging from mild to severe i.e. more than 5

Exclusion Criteria:

* Patients with hypoventilation syndrome
* Patients with chronic obstructive pulmonary disease
* Patients who have unstable hemodynamic state, who experienced intolerance to HFNC or CPAP
* Patients who are pregnant
* Patients recently underwent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Apnea/Hypopnea Index count using High Flow Nasal Cannula oxygen device and Continuous Positive Pressure Airway device on patients with Obstructive Sleep Apnea | two nights
  the Apnea/Hypopnea Index (AHI) is 5 events or less
Sleep architecture while using High Flow Nasal Cannula oxygen device | two nights
  Standard sleep architecture: sleep breathing disorder e.g. apnea, hypopnea, snoring Oxygenation : minimum oxygen saturation, duration of desaturation and number of desaturation Arousals : number and index
Tolerance and acceptability of High Flow Nasal Cannula by patients compared to the standard Continuous Positive Airway Pressure | two nights
  Comparison of High Flow Nasal Cannula device compared to the Continuous Positive Airway Pressure for a long term usage; being assessed in
  1. How well did you accept the device yesterday?
  2. How comfortable was the usage of the device?
  3. Was the used mask comfortable? (1)not acceptable, (2)tolerable, (3)acceptable, (4)well received, (5)excellent
  4. Did you face any difficulties breathing through your nose while using the device last night?
  5. Did you have any of these symptoms while using the mask last night? Nasal dryness, Mouth dryness, Runny nose, Fear or anxiety, Congested nose
  6. Did you feel any air leakage from the mask last night ?
  7. Was it hard keeping the mask on while sleeping?
  8. Are you prepared to use the CPAP machine as a therapy daily?

SECONDARY OUTCOMES:
Changes in sleep structure compared to the diagnostic night | two night
  Refine the sleep structure with the usage of the device, the count of Apnea/Hypopnea index, number of arousals, number of desaturations

CONTACTS AND LOCATIONS:
Overall Officials: Siraj O Wali, Professor, Study Director — Teaching Assistant at King Abdulaziz University
Locations (1):
- King Abdulaziz University Hospital, Jeddah, Western, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
The study outcome might be shared as well as the methodology

REFERENCES:
- [Derived] Wali S, Batawi G, Bin Afeef G, Bamagoos AA, Jamal A, Kanbr O, Alshumrani R, Alhejaili F, Badr MS. The effectiveness of high-flow nasal cannula therapy in comparison with continuous positive airway pressure therapy in patients with obstructive sleep apnea: an open-label randomized crossover trial. J Clin Sleep Med. 2025 Jun 1;21(6):1023-1031. doi: 10.5664/jcsm.11640. PMID 40051198